CLINICAL TRIAL: NCT07391657
Title: A Phase III Open-label, Randomised, Multicentre Study Comparing AZD0120, a Dual-Targeting Autologous Chimeric Antigen Receptor T-cell (CART) Therapy Directed Against BCMA and CD19, Versus Standard Regimens in Participants With Relapsed Refractory Multiple Myeloma.
Brief Title: A Phase III, Open-label, Randomised, Multicentre Study to Evaluate AZD0120 in Participants With Relapsed Refractory Multiple Myeloma.
Acronym: DURGA-4
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8311C00001; AZD0120 (Other: AstraZeneca)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Refractory Multiple Myeloma
Keywords: BCMA; CAR-T; CD19
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; carfilzomib; Dexamethasone; Bortezomib; pomalidomide

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): AZD0120
  Interventions: Biological: AZD0120
- Arm B (Active Comparator): 1 of the following 4 standard regimens per investigator choice; DKd, DPd, PVd, Kd.
  Interventions: Drug: Daratumumab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Bortezomib; Drug: Pomalidomide

INTERVENTIONS:
Biological: AZD0120 — CAR-T Cells
  Arms: Arm A
Drug: Daratumumab — Daratumumab
  Other Names: Darzalex
  Arms: Arm B
Drug: Carfilzomib — Carfilzomib
  Other Names: Kyprolis
  Arms: Arm B
Drug: Dexamethasone — Dexamethasone
  Arms: Arm B
Drug: Bortezomib — Bortezomib
  Other Names: Velcade
  Arms: Arm B
Drug: Pomalidomide — Pomalidomides
  Other Names: Pomalyst and Imnovid
  Arms: Arm B

SUMMARY:
This is a randomised, multicentre, controlled, open-label, Phase III global study comparing the efficacy and safety of AZD0120 versus standard regimens (DKd [daratumumab, carfilzomib, and dexamethasone], DPd [daratumumab, pomalidomide, and dexamethasone], PVd [pomalidomide, bortezomib and dexamethasone], or Kd [carfilzomib and dexamethasone]) in participants with RRMM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Documented diagnosis of multiple myeloma according to the IMWG diagnostic criteria
* Documented evidence of measurable disease:

  1. Serum M-protein level ≥ 1 g/dL
  2. Urine M-protein level ≥ 200 mg/24h
  3. Serum immunoglobulin free light chain ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Documented evidence of PD by IMWG 2016 criteria based on investigator's determination during or after the most recent line of therapy. Participants with only 1 prior line of therapy must have progressed within 47 months of a stem cell transplant, or if not transplanted, then within 42 months of starting initial therapy
* Received 1 to 3 lines of prior therapy including an IMiD and either a PI or a CD38 antibody. Participant must have undergone at least 2 complete cycles of treatment for each line of therapy, unless PD was the best response to the line of therapy
* Eligible to receive at least one of the standard regimens (DKd, PVd, DPd, or Kd) as determined by the Investigator.
* ECOG performance status score of 0 to 1
* Adequate hematology and chemistry laboratory values:

  1. Haemoglobin ≥ 8.0 g/dL
  2. Absolute neutrophil count ≥ 1 × 10^9/L (1000 per mm3)
  3. Platelet count ≥ 75 × 10^9/L (75000 per mm3) in participants with < 50% of bone marrow nucleated cells are plasma cells or ≥ 50 × 10^9/L (50000 per mm3) in participants with ≥ 50% of bone marrow nucleated cells are plasma cells
  4. Absolute lymphocyte count ≥ 300/µL (0.3 × 109/L)
  5. Total bilirubin ≤ 1.5 × ULN in the absence of Gilbert's syndrome or ≤ 3 × ULN if the participant has Gilbert's syndrome. AST and ALT≤ 3.0 × ULN. CrCl by Cockcroft and Gault method ≥ 30 mL/minute

Exclusion Criteria:

* Known active, or prior history of CNS involvement or exhibits clinical signs of meningeal involvement of MM.
* Primary amyloidosis, active plasma cell leukaemia, Waldenstrom macroglobulinemia or Polyneuropathy Organomegaly Endocrinopathy M-protein and Skin (POEMS) syndrome.
* Participants with primary refractory MM (failed to generate at least a minimal response to any prior therapy)
* Significant neurological or psychiatric condition
* Significant medical condition that places the participant at an unacceptable risk for treatment-related complications
* Previously received any prior BCMA-targeted treatment
* Previously received CAR-T or CAR-NK therapy directed at any target
* Previously received T-cell engager therapy directed at any target
* Previously received allogeneic stem cell transplantation at any time during prior therapy or received autologous stem cell transplantation within 12 weeks of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the superiority of AZD0120 relative to standard therapy (DKd, DPd, PVd, or Kd) by assessment of PFS in participants with RRMM. | 3 years
  PFS: defined as time from randomisation until progression according to IMWG 2016 criteria as assessed by BICR, or death due to any cause, whichever occurs first.
To demonstrate the superiority of AZD0120 relative to standard therapy (DKd, DPd, PVd, or Kd) by assessment of MRD negativity rate at 9 months in participants with RRMM. | 2 years
  MRD negative CR rate at 9 months: defined as the proportion of participants with MRD negative status and have a response of CR or sCR (according to the IMWG 2016 criteria) at 9 months (± 3 months) from randomisation before initiation of subsequent anti-myeloma therapy.

SECONDARY OUTCOMES:
To further demonstrate the effectiveness of AZD0120 relative to standard therapy (DKd, DPd, PVd, or Kd) by assessment of CRR in participants with RRMM. | 2 years
To further demonstrate the effectiveness of AZD0120 relative to standard therapy (DKd, DPd, PVd, or Kd) by assessment of ORR in participants with RRMM. | 2 years
To further demonstrate the effectiveness of AZD0120 relative to standard therapy (DKd, DPd, PVd, or Kd) by assessment of OS in participants with RRMM. | 5 years

CONTACTS AND LOCATIONS:
Locations (94):
- United States (37):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Santa Monica, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Australia (6):
  - Research Site, Camperdown
  - Research Site, Darlinghurst
  - Research Site, Fitzroy
  - Research Site, Liverpool
  - Research Site, Melbourne
  - Research Site, Murdoch
- Brazil (2):
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (6):
  - Research Site, Lille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Toulouse
- Germany (10):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Nuremberg
  - Research Site, Würzburg
- Italy (5):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Rozzano
  - Research Site, Torino
- Japan (6):
  - Research Site, Bunkyō City
  - Research Site, Kashiwa
  - Research Site, Kyoto
  - Research Site, Nagoya
  - Research Site, Shibuya-ku
  - Research Site, Shinjuku-ku
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Valencia
- Research Site, Taipei, Taiwan
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Bristol
  - Research Site, Glasgow, Scotland
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/